CLINICAL TRIAL: NCT02072525
Title: A Protocol to Collect Human Serum Samples From Healthy Adults
Brief Title: A Protocol to Collect Human Serum Samples From Healthy Adults for Use as Quality Controls Samples in GlaxoSmithKline (GSK) Biologicals' Assays
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 200612
Record Dates: First submitted 2014-02-20; First posted 2014-02-26 (Estimated); Last update posted 2017-11-27 (Actual); Status verified 2017-11

CONDITIONS: Meningococcal
Keywords: Pertussis; Healthy adults; Tetanus; Human serum samples; Streptococcus; Diphtheria; Plasma; Meningococcus
MeSH Terms: conditions — Whooping Cough; Tetanus; Diphtheria | interventions — Meningococcal Vaccines; Boostrix; 23-valent pneumococcal capsular polysaccharide vaccine; 13-valent pneumococcal vaccine

ARMS (9):
- Mtdap1 Group (Experimental): Subjects will receive concomitant doses of Menveo and Boostrix.
  Interventions: Biological: Menveo®; Biological: Boostrix®
- Mtdap2 Group (Experimental): Subjects will receive concomitant doses of Menveo and Boostrix.
  Interventions: Biological: Menveo®; Biological: Boostrix®
- Mtdap3 Group (Experimental): Subjects will receive concomitant doses of Menveo and Boostrix.
  Interventions: Biological: Menveo®; Biological: Boostrix®
- Pneum1 Group (Experimental): Subjects will receive a dose of Pneumovax 23.
  Interventions: Biological: Pneumovax 23®
- Pneum2 Group (Experimental): Subjects will receive a dose of Pneumovax 23.
  Interventions: Biological: Pneumovax 23®
- Pneum 3 Group (Experimental): Subjects will receive a dose of Pneumovax 23.
  Interventions: Biological: Pneumovax 23®
- Prev1 Group (Experimental): Subjects will receive a dose of Prevnar 13.
  Interventions: Biological: Prevnar 13®
- Prev2 Group (Experimental): Subjects will receive a dose of Prevnar 13.
  Interventions: Biological: Prevnar 13®
- Prev3 Group (Experimental): Subjects will receive a dose of Prevnar 13.
  Interventions: Biological: Prevnar 13®

INTERVENTIONS:
Biological: Menveo® — One dose administered intramuscularly (IM) in the upper left deltoid of the arm.
  Arms: Mtdap1 Group; Mtdap2 Group; Mtdap3 Group
Biological: Boostrix® — One dose administered intramuscularly (IM) in the upper right deltoid of the arm.
  Arms: Mtdap1 Group; Mtdap2 Group; Mtdap3 Group
Biological: Pneumovax 23® — One dose administered intramuscularly (IM) in the non-dominant deltoid of the arm.
  Arms: Pneum 3 Group; Pneum1 Group; Pneum2 Group
Biological: Prevnar 13® — One dose administered intramuscularly (IM) in the non-dominant deltoid of the arm.
  Arms: Prev1 Group; Prev2 Group; Prev3 Group

SUMMARY:
The purpose of this study is to collect serum samples for use as quality control samples in GSK assays. The serum samples need to include samples with low, medium and high antibody titers/concentrations, which cover the assay range.

DETAILED DESCRIPTION:
The purpose of this protocol is to source human serum from plasma from healthy adults for use as control samples in the assays supporting the clinical development of GSK Biologicals' vaccines for the prevention of invasive infections caused by Neisseria meningitidis, Streptococcus pneumoniae, Corynebacterium diphtheriae, Clostridium tetani and Bordetella pertussis. At the final visit, a small volume of whole blood will be obtained in addition to plasma, to allow for head to head comparison of serum obtained from whole blood (off-clot serum) and from plasma (serum derived from re-calcified plasma). In addition, sera generated in this clinical trial could potentially be used as control samples for other vaccine programs to help assure the quality of the analytical methods.

Subjects 18 through 49 years of age (have not yet achieved 50th birthday) will be randomized to receive Menveo + Boostrix and subjects 50 to 55 years of age will be randomized to receive either Pneumovax 23 or Prevnar 13 and will serve as donors of human serum in this study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
* A male or female between, and including, 18 and 55 years of age at the time of the first vaccination.
* Written informed consent obtained from the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study, with no medical conditions that in the opinion of the investigator prevents the subject from participating in the study.
* Subjects must weigh at least 110 pounds (50 kg).
* Female subjects of non-childbearing potential may be enrolled in the study.

  * Non-childbearing potential is defined as pre-menarche, current tubal ligation, hysterectomy, ovariectomy or post-menopause.
* Female subjects of childbearing potential may be enrolled in the study, if the subject:

  * has practiced adequate contraception for at least 30 days prior to vaccination, and
  * has a negative pregnancy test on the day of vaccination, and
  * has agreed to continue adequate contraception for the entire duration of the subject's participation in the trial.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) within 30 days preceding the dose of study vaccine, or planned use during the study period.
* Subjects seropositive for hepatitis B surface antigen (HBsAg), antibody to hepatitis C virus (anti-HCV) or HIV.
* Chronic administration (defined as more than 14 days in total) of immunosuppressants or other immune-modifying drugs within six months prior to the vaccine dose. Inhaled and topical steroids are allowed.
* Administration of long-acting immune-modifying drugs at any time during the study period.
* Any antibiotic taken during the period from 14 days before the collection of plasma up to the day of collection of plasma.
* Any medication based on methyl phenidate HCL such as Metadate® or Concerta® or other CNS stimulants used to treat attention-deficit disorder or attention-deficit hyperactivity disorder taken during the period of 14 days before the collection of plasma up to the day of collection of plasma.
* Subjects who donated >500 mLs of blood within 60 days prior to any plasma collection visits (plasmapheresis).
* Subjects who lost >200 mL of red blood cells during a single apheresis procedure or lost red blood cells on more than one occasion during apheresis within the previous 60 days.
* Ongoing anemia as indicated by either (i) hemoglobin values, (ii) serum ferritin, or (iii) hematocrit values below the lower limit of the laboratory-specified reference range. If the laboratory results demonstrate an anemia, no further protocol procedures will be performed, and the subject will be referred for appropriate medical management. The subject may participate in this study following therapy and evidence that the anemia has been resolved.
* Bleeding disorder and/or a clinical laboratory platelet count value below the lower limit of the laboratory-specified reference range.
* Planned administration/administration of a vaccine not foreseen by the study protocol within the period starting 30 days before and 30 days after the dose of vaccine, with the exception of licensed inactivated influenza vaccine.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational vaccine/product.
* Family history of congenital or hereditary immunodeficiency.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine(s).
* Hypersensitivity to latex.
* Serious chronic illness.
* Acute disease and/or fever at the time of vaccination (Day 0).

  * Fever is defined as temperature ≥ 37.5°C /99.5°F for oral, axillary or tympanic route, or ≥ 38.0°C /100.4°F on rectal route. The preferred route for recording temperature in this study will be oral.
  * Subjects with a minor illness (such as mild diarrhoea, mild upper respiratory infection) without fever may, be enrolled at the discretion of the investigator.
* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory screening tests.
* History of chronic alcohol consumption and/or drug abuse.
* Administration of immunoglobulins and/or any blood products within the 3 months preceding the first dose of study vaccine or planned administration during the study period.
* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions.
* Any confirmed or suspected immunosuppressive or immunodeficient condition (congenital or secondary) based on medical history and history directed physical examination (no laboratory testing at the screening visit is required).

Additional exclusion criteria for subjects 18-49 years of age

* Previous vaccination against diphtheria and/or tetanus within the past 5 years and/or Neisseria meningitidis since birth.
* Progressive neurological disorders, including uncontrolled epilepsy or progressive encephalopathy.
* Subjects who have experienced an encephalopathy of unknown etiology, occurring within 7 days following previous vaccination with a pertussis containing vaccine.
* Subjects who have experienced transient thrombocytopenia or neurological complications following an earlier immunization against diphtheria and/or tetanus.
* If any of the following events had occurred in temporal relation to previous administration of whole-cell DTP or acellular DTP vaccine:

  * Temperature of ≥ 40.0°C within 48 hours of vaccination, not due to another identifiable cause.
  * Collapse or shock like state (hypotonic hyporesponsive episode) within 48 hours of vaccination.
  * Persistent, inconsolable crying lasting ≥ 3 hours, occurring within 48 hours of vaccination.
  * Convulsions with or without fever, occurring within 3 days of vaccination.

Additional exclusions criterion for subjects 50-55 years of age

• Previous vaccination against Streptococcus pneumoniae.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 359 (Actual)
Dates: Start 2014-04-01 (Actual); Primary Completion 2015-06-02 (Actual); Study Completion 2015-06-02 (Actual)

PRIMARY OUTCOMES:
Collection of human plasma for conversion into serum. | At Visit 2 (Day 0).
  Collection of human plasma for conversion into serum for use as control samples in GSK Biologicals' assays in support of Neisseria meningitidis, Streptococcus pneumoniae, Corynebacterium diphtheriae, Clostridium tetani and Bordetella pertussis vaccine development programs.
Collection of human plasma for conversion into serum. | At 10 days post-vaccination.
  Collection of human plasma for conversion into serum for use as control samples in GSK Biologicals' assays in support of Neisseria meningitidis, Streptococcus pneumoniae, Corynebacterium diphtheriae, Clostridium tetani and Bordetella pertussis vaccine development programs.
Collection of human plasma for conversion into serum. | At 30 days post-vaccination.
  Collection of human plasma for conversion into serum for use as control samples in GSK Biologicals' assays in support of Neisseria meningitidis, Streptococcus pneumoniae, Corynebacterium diphtheriae, Clostridium tetani and Bordetella pertussis vaccine development programs.
Collection of human plasma for conversion into serum. | At 60 days post-vaccination.
  Collection of human plasma for conversion into serum for use as control samples in GSK Biologicals' assays in support of Neisseria meningitidis, Streptococcus pneumoniae, Corynebacterium diphtheriae, Clostridium tetani and Bordetella pertussis vaccine development programs.
Collection of human plasma for conversion into serum. | At 120 days post-vaccination
  Collection of human plasma for conversion into serum for use as control samples in GSK Biologicals' assays in support of Neisseria meningitidis, Streptococcus pneumoniae, Corynebacterium diphtheriae, Clostridium tetani and Bordetella pertussis vaccine development programs.

SECONDARY OUTCOMES:
Occurrence of serious adverse events related to vaccination and to lack of vaccine efficacy throughout the study. | Throughout the study (Day 0 to Day 30 - Day 180).

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Sherbrooke, Quebec, Canada

REFERENCES:
- See also: GSK-CSR CTRS PDF link given. — https://www.gsk-clinicalstudyregister.com/files2/200612%20-%20Clinical-Study-Result-Summary.pdf